CLINICAL TRIAL: NCT05011292
Title: Strengthening and Supporting the Diabetes Early Prevention Efforts of Pediatric Primary Healthcare Providers
Brief Title: Well-child Visit Video Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jean Welsh, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001393; P30DK111024 (NIH)
Record Dates: First submitted 2021-08-13; First posted 2021-08-18 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes
Keywords: Prevention; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group includes parents that will view an educational video about a topic other than infant SCB consumption.
  Interventions: Behavioral: Survey on child feeding and related knowledge and practices; Behavioral: Educational Video other than SCB
- Intervention Group (Experimental): The intervention group will include those parents who participate in the study after the control data has been collected and two SCB reduction-related videos have been introduced (one for showing at the 4-month visit and one for the 12-month visit).
  Interventions: Behavioral: Educational Video about SCB; Behavioral: Survey on child feeding and related knowledge and practices

INTERVENTIONS:
Behavioral: Educational Video about SCB — 3-4 minutes video about SCB.
  Arms: Intervention Group
Behavioral: Survey on child feeding and related knowledge and practices — Short survey about infant feeding practices (3-4 minutes). No identifying information will be collected. The general scope of topics covered in the surveys will be attitudes toward the sugar-containing beverage reduction (SCB) videos played at the clinic as well as SCB knowledge and practices of parents and their children.
Behavioral: Educational Video other than SCB — Educational video about a topic other than infant SCB consumption.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine if incorporating videos on the importance of minimizing infant sugar-containing beverage (SCB) consumption into well-child visit protocols increases parents' SCB-related knowledge and their compliance with related early feeding recommendations. The study also aims to determine whether these videos increase the frequency and quality of the SCB-related reduction education and counseling provided to parents during well-child visits.

DETAILED DESCRIPTION:
The purpose of this study is to determine if incorporating videos on the importance of minimizing infant sugar-containing beverage (SCB) consumption into well-child visit protocols increases parents' SCB-related knowledge and their compliance with related early feeding recommendations. The study also aims to determine whether these videos increase the frequency and quality of the SCB-related reduction education and counseling provided to parents during well-child visits.

The populations to be studied include:

1. Parents of children attending a 4, 6, 9, 12 or 15-month well-child visit (Main study)
2. A subsample of parents from above that agree to complete a baseline and follow-up knowledge and practice survey 5 to 6 months after enrollment. (Long-Term follow-up study)
3. Members of the clinic team who participate in the project (Key informant interviews)

Participants in the main study will include parents attending a 4-month, 6-month, 9-month, 12-month or 15-month well-child visit at Hughes Spalding clinic, Atlanta GA. During their 4-month or 12-month clinic visit, parents will be offered to view a video (3 minutes) and complete a short survey about it afterwards (2 minutes). Parents attending their child's 6, 9 or 15-month well-child visit will be asked to complete a short survey about infant feeding practices (3-4 minutes). No identifying information will be collected. A waiver of consent is being requested for this component of the study.

A subsample of the parents referenced above will be invited by co-investigators on the clinic team to participate in a long-term follow-up survey to assess the extent to which viewing the well-child visit videos has an impact of knowledge and/or behavior that is sustained. Those who consent will be asked to provide their first name and email address in order to enable the follow up survey to be completed on-line. No other PHI will be collected. A study ID will be assigned and only the PI and the statistician will have access to the code that links identifiers to subjects. Sub sample participants will be asked to view a video at the child's 4-month or 12-month well-child visit, to complete a survey assessing their response to the video as well as their infant feeding practices. This survey will be repeated during their 6-month or 15-month well-child visit and again, by email, 2 to 3 months later. Total participation time is expected to be <20 minutes.

Key informant interviews will be completed by members of the clinic team involved in the various aspects of the study. These will be done as time allows and will involved discussions of 5 to 30 minutes depending on the availability of the staff members. No identifying information will be collected as part of these interviews.

The general scope of topics covered in the surveys and key informant interviews will be attitudes toward the sugar-containing beverage reduction (SCB) videos played at the clinic as well as SCB knowledge and practices of parents and their children. Participant burden for parents will range from about 6 minutes for those completing only the initial survey to an estimated 20 minutes for the sub-sample of parents involved in the long-term follow-up. Clinic staff that are involved in the key informant interviews will spend 5-30 minutes participating in the study.

Willingness to participate in the long-term follow-up study will be assessed by clinic staff/study co-investigators who will complete an informed consent process (waiver of written consent requested) for those interested. The only identifiable information collected will be a participants name and phone number.

PHI will be forwarded in encrypted emails to the research team using a secure Children's Healthcare of Atlanta email account and entered into a password protected RedCap database. Survey data will also be collected and stored in that same database. Data confidentiality will be assured by using ID numbers for those who provide identifiable contact information (name and phone number). The code that links identifiers to subjects will be stored on locked and password protected devices, with access only give to study staff who need the information to perform the study.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age, AND
* Being a parent/caregiver of a child age 4-15 months, AND
* Attending a well-child visit at the collaborating pediatric primary care clinic and planning to continue during the pilot implementation.

Exclusion Criteria:

* Parents/caregivers with cognitive or behavioral limitations that preclude completion of the survey
* Parents/caregivers of children with conditions that require special feeding protocols, e.g. tube feedings, high calorie supplements
* Parent/caregivers who are not able to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Welsh, PhD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta - Hughes Spalding Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: The control group includes parents that will view an educational video and respond to survey questions about a topic other than infant SCB consumption (4 or 12-month well-child visit) or complete an infant feeding assessment survey (6-, or 15-month well-child visit).
- Intervention Group: The intervention group includes parents that view a SCB-reduction video while attending their child's 4-month or 12-month well-child visit.
- Clinical Staff: Clinical Staff providing the video to the study participants during clinic operations were asked to answer a few written and verbal questions regarding the well-child visit videos presented in the clinic.
Period: Overall Study
Arm/Group | Control Group | Intervention Group | Clinical Staff
Started | 116 | 267 | 5
Completed | 116 | 56 | 5
Not Completed | 0 | 211 | 0

BASELINE CHARACTERISTICS:
Population: Data was not collected for the Clinical Staff group.
Groups:
- Control Group: The control group includes parents that will view an educational video about a topic other than infant SCB consumption (4 or 12-month well-child visit) and respond to survey questions or complete an infant feeding assessment survey (6, or 15-month well-child visit).
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention Group | Clinical Staff | Total
Number analyzed (Participants) | 116 | 267 | 0 | 383
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 85 | 213 |  | 298
  >=65 years | 31 | 54 |  | 85
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 231 |  | 335
  Male | 12 | 36 |  | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 |  | 15
  Not Hispanic or Latino | 110 | 258 |  | 368
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 105 | 238 |  | 343
  White | 10 | 27 |  | 37
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 1 | 2 |  | 3
Region of Enrollment [Number; unit: participants]
  United States | 116 | 267 |  | 383
Number of participants that viewed and completed survey on perceptions of educational video [Count of Participants; unit: Participants] | 62 | 267 |  | 329
Number of participants that completed and infant feeding practices survey [Count of Participants; unit: Participants] | 54 | 267 |  | 321

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Parents Who Are Aware of Infant Fruit Juice Consumption Recommendations
Description: This will be assessed by asking parents if they are "aware of any expert recommendations related to the age or amount of fruit juice given to infants and/or young children?". Those responding "yes" will be asked to specify the recommendation. If their response is correct, they will be recorded as knowledgeable.
Time Frame: 0-3 months post-intervention
Population: For the control Group: Include participants that complete the fruit juice recommendation question on the infant feeding assessment survey.
  For the Intervention Group: Includes only those who viewed the intervention video at their child's 4-month or 12-month well child visit and who attend their 6-month or 15-month well-child visit and complete the fruit juice recommendation question on the infant feeding survey.
Measure: Number; unit: percentage of participants
Groups:
- Control Group: The control group includes parents that will view an educational video about a topic other than infant SCB consumption (4 or 12-month well-child visit) or complete an infant feeding assessment survey (6, or 15-month well-child visit).
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 46 | 44
percentage of participants | 19.57 | 27.27

2. Primary Outcome: Percentage of Parents Who Report That They do Not Give Their Young Children Fruit Juice
Description: Parents will be asked if they give their young child fruit juice. Response options will be "yes" or "no". Participants responding "no" are reported.
Time Frame: 2-3 months post-intervention
Population: For the Control group: parents attending their child's 6-month well-child visit and responding to the survey question about their child's fruit consumption.
  For the Intervention Group: Participants include those that viewed a video at the 4-month visit, attend the 6-month visit, and respond to the survey question about their child's fruit juice consumption.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 36 | 38
percentage of participants | 58.3 | 60.5

3. Primary Outcome: Percentage of Parents Who Report That They do Not Give Their Young Children Sugar-sweetened Beverages.
Description: Parents will be asked if they give their young child sugar-sweetened beverages. Response options will be "yes" or "no". Percentage of parents who report"no" will be reported.
Time Frame: 2-3 months post-intervention
Population: For the Control Group: Includes parents of participants attending their child's 15-month well-child visit and responding to the survey question about their child's sugar-sweetened beverage consumption.
  For the Intervention Group: Participants include those that viewed a video at the 12-month visit, attend the 15-month visit, and respond to the survey question about their child's sugar-sweetened beverage consumption.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 12 | 9
percentage of participants | 8.3 | 55.6

4. Secondary Outcome: Percentage of Clinic Staff Who Report That the SCB Consumption Related Videos Were Easy to Incorporate Into the Flow of Clinic Operations
Description: This outcome will be assessed with the key informant survey that specifically asks if staff found it "easy to integrate the videos into the flow of clinic operations". Positive responses will be reported.
Time Frame: Up to 9 months post-intervention
Measure: Number; unit: percentage of participants
Groups:
- Clinical Staff: Clinical Staff providing the video to the study participants during clinic operations will be asked to answer a few written and verbal questions regarding the well-child visit videos presented in the clinic.
Arm/Group | Clinical Staff
Number analyzed (Participants) | 5
percentage of participants | 80

5. Secondary Outcome: Percentage of Parents Who Viewed an Intervention Video Report That They Enjoyed it
Description: Parents will be asked specifically if they "enjoyed the video". Responses will be on a 5-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree".
  Percentage of parents who "agree" or "strongly agree" are reported.
Time Frame: immediately post-intervention, within 30 minutes
Population: The Intervention Group includes participants that viewed a video at their child's 4-month or 12-month visit.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 62 | 267
percentage of participants | 87 | 95.9

6. Secondary Outcome: Percentage of Parents Who Viewed an Intervention Video Report That They Learned Something From it
Description: Parents will be asked specifically if they "learned something" from it. Responses will be on a 5-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree".
  Percentage of parents who "agree" or "strongly agree" are reported.
Time Frame: immediately post-intervention, within 30 minutes
Population: The Control Group includes participants attending the child's 4-month or 12-month well-child visit.
  The Intervention Group includes participants that viewed a video at their child's 4-month or 12-month visit.
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Intervention Group
Number analyzed (Participants) | 62 | 267
percentage of participants | 83.9 | 95.5

ADVERSE EVENTS:
Time Frame: During follow up time (up to 12 months post intervention).
Description: Adverse event data was not collected for the Clinical Staff participants.
Arm/Group | Control Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/267
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/267
Other Adverse Events (participants affected / at risk) | 0/116 | 0/267

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT05011292/Prot_SAP_001.pdf
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT05011292/ICF_000.pdf